CLINICAL TRIAL: NCT03315299
Title: Individual Patient Expanded Access for Use of Gilteritinib (ASP2215) for Patient Y.A.
Brief Title: Individual Patient Expanded Access Gilteritinib (ASP2215)
Status: No longer available | Type: Expanded Access
Sponsor: Etan Orgel (Other)
Collaborators: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Etan Orgel, Principal Investigator, Children's Hospital Los Angeles
Organization: Children's Hospital Los Angeles (Other)
Other Study IDs: CHLA-17-00428
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: AML
MeSH Terms: interventions — gilteritinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: ASP2215 — Subject will take ASP2215 by mouth daily for 28 day cycles
  Other Names: gilteritinib

SUMMARY:
The purpose of this study is to provide expanded access to ASP2215 for a single subject with refractory FLT3-mutated AML without access to comparable or alternative therapy.

DETAILED DESCRIPTION:
This treatment protocol is being conducted in a single pediatric patient while phase 3 ASP2215 studies are ongoing in adult subjects with FLT3-mutated AML.

The subjects will enter the screening period up to 2 weeks prior to the start of treatment.

The subject will be administered treatment over 28-day cycles.

The subjects will complete visits on cycle 1 days 1, 4, 8, 15; cycle 2 days 1, 15, and day 1 of each cycle thereafter until discontinued from the study for toxicity, disease progression, or lack of continued benefit in the judgement of the investigator.

An end of treatment visit will be performed within 7 days after last dose of the investigation product (ASP2215), or prior to initiation of another anticancer therapy, whichever occurs earlier, followed by a 30-day follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Institutional Review Board-/Independent Ethics Committee-approved written Informed Consent and privacy language as per national regulation (e.g., Health Insurance Portability and Accountability Act authorization for United States sites) must be obtained from the subject or legally authorized representative prior to any study-related procedures (including withdrawal of prohibited medication, if applicable).
2. Subject has a diagnosis of primary AML or AML secondary to myelodysplastic syndrome (MDS) or therapy-related AML according to World Health Organization classification [Swerdlow et al., 2008] as determined by pathology review at the treating institution.
3. Subject has presence of the FLT3 mutation (internal tandem duplication [ITD] and/or tyrosine kinase domain [TKD] [D835/I836] mutation) in bone marrow or peripheral blood as determined by local laboratory.
4. Subject has refractory or relapsed AML (with or without hematopoietic stem cell transplant [HSCT]) or AML in complete remission (CR) with minimal residual disease by flow cytometry or genetic testing after induction/consolidation regimen.
5. In the judgment of the investigator, there is no comparable or satisfactory alternative therapy to treat the subject's AML.
6. Subject has not received any chemotherapy or investigational agent within at least 5 half-lives after stopping that drug and before starting gilteritinib.
7. Subject must meet the following criteria as indicated on clinical laboratory tests:

   * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x institutional upper limit of normal (ULN)
   * Serum total bilirubin < 2.5 mg/dL, except for subjects with Gilbert's syndrome
   * Serum potassium and serum magnesium > institutional lower limit of normal (LLN).
8. Subject is able to tolerate oral administration of study drug.
9. Subject who has developed overall grades II-IV graft-versus-host disease (GVHD) must satisfy the following criteria:

   * No requirement of > 0.5 mg/kg of prednisone (or equivalent) daily dose within 1 week of randomization
   * No escalation of immunosuppression in terms of increase of corticosteroids or addition of new agent / modality in prior 2 weeks (note that increasing calcineurin inhibitors or sirolimus to achieve therapeutic trough levels is allowed).
10. Female subject must either:

    * Be of nonchildbearing potential:
    * Postmenopausal (defined as at least 1 year without any menses) prior to screening, or
    * Documented surgically sterile or status posthysterectomy (at least 1 month prior to screening)
    * Or, if of childbearing potential,
    * Agree not to try to become pregnant during the study and for 180 days after the final study drug administration
    * And have a negative urine pregnancy test at screening
    * And, if heterosexually active, agree to use consistently 2 forms of effective contraception per locally accepted standards (1 of which must be a barrier method) starting at screening and throughout the study period and for 180 days after the final study drug administration.
11. Female subject must agree not to breastfeed or donate ova starting at screening and throughout the study period, and for 180 days after the final study drug administration.
12. Subject agrees not to participate in another interventional study while on treatment.
13. Subject who has a diagnosis of human immunodeficiency virus (HIV) may be enrolled as long as their disease is under control on antiretroviral therapy. Precautions should be taken to modify their highly active antiretroviral therapy (HAART) regimen to minimize drug interactions.

Exclusion Criteria:

Subject will be excluded from participation if any of the following apply:

1. Subject is eligible for enrollment in another ongoing clinical study of gilteritinib.
2. Subject has participated in a previous or ongoing open-label, randomized treatment study of gilteritinib.
3. Subject with Fridericia-corrected QT interval (QTcF) > 450 ms at screening based on local reading.
4. Subject with Long QT Syndrome at screening.
5. Subject was diagnosed as acute promyelocytic leukemia (APL).
6. Subject has BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
7. Subject has clinically significant coagulation abnormality unless secondary to AML in the opinion of the investigator.
8. Subject has active hepatitis B or C or an active hepatic disorder.
9. Subject has uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia, or New York Heart Association (NYHA) Class IV heart failure.
10. Subject requires treatment with concomitant drugs that are strong inducers of CYP3A.
11. Subject requires treatment with concomitant drugs that are strong inhibitors or inducers of P-gp with the exception of drugs that are considered absolutely essential for the care of the subject.
12. Subject requires treatment with concomitant drugs that target serotonin 5HT1R or 5HT2BR or sigma nonspecific receptor with the exception of drugs that are considered absolutely essential for the care of the subject.
13. Subject has any condition which, in the investigator's opinion, makes the subject unsuitable for study participation.

Ages: 12 Years to 15 Years | Sex: Female
Age Groups: Child
Gender Based: Yes — Single patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States